CLINICAL TRIAL: NCT06855576
Title: A Phase I, Randomised, Open Label, Single Center, Single Oral Dose, Three Treatment, Three Period, Three Sequence, Change-over Bioequivalence Study of Paracetamol Orodispersible Tablet 500 mg (Haleon) to Assess Bioequivalence With Alvedon 500 mg Film-Coated Tablet (Haleon, Sweden) and Panadol 500 mg Film-Coated Tablet (Haleon, Australia) in Healthy Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Paracetamol With Oral Single Dose Administration in Healthy Adult Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 300141; 2024-514198-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-28; First posted 2025-03-04 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Fever; Pain
MeSH Terms: conditions — Fever; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Product (Experimental): Participants will be randomly assigned as per cross-over design to receive oral administration of one paracetamol ODT (test product) on day 1 of period 1, one Alvedon film-coated tablet (reference product 1) on day 1 of period 2 and one Panadol film-coated tablet (reference product 2) on day 1 of period 3, each under fasting conditions. There will be at least 72 hours of washout between each period (no more than 7 days).
  Interventions: Drug: Paracetamol ODT; Drug: Alvedon film-coated tablet; Drug: Panadol film-coated Tablet
- Reference Product 1 (Active Comparator): Participants will be randomly assigned as per cross-over design to receive oral administration of one Alvedon film-coated tablet (reference product 1) on day 1 of period 1, one Panadol film-coated tablet (reference product 2) on day 1 of period 2 and one paracetamol ODT (test product) on day 1 of period 3, each under fasting conditions. There will be at least 72 hours of washout between each period (no more than 7 days).
  Interventions: Drug: Paracetamol ODT; Drug: Alvedon film-coated tablet; Drug: Panadol film-coated Tablet
- Reference Product 2 (Active Comparator): Participants will be randomly assigned as per cross-over design to receive oral administration of one Panadol film-coated tablet (reference product 2) on day 1 of period 1, and one paracetamol ODT (test product) on day 1 of period 2 and one Alvedon film-coated tablet (reference product 1) on day 1 of period 3, each under fasting conditions. There will be at least 72 hours of washout between each period (no more than 7 days).
  Interventions: Drug: Paracetamol ODT; Drug: Alvedon film-coated tablet; Drug: Panadol film-coated Tablet

INTERVENTIONS:
Drug: Paracetamol ODT — Experimental Paracetamol 500 mg ODT
Drug: Alvedon film-coated tablet — Marketed Paracetamol 500 mg film-coated tablet
Drug: Panadol film-coated Tablet — Marketed Paracetamol 500 mg film-coated tablet

SUMMARY:
This study aims to evaluate the bioequivalence of new formulated orodispersible tablet (ODT) containing 500 milligram (mg) paracetamol in comparison to the European marketed Alvedon (paracetamol) 500 mg film-coated tablets and the Australian marketed Panadol (paracetamol) 500 mg film-coated tablets as reference products.

DETAILED DESCRIPTION:
This will be a single center, open-label, randomized (order of treatments), balanced, 3-period, 3-sequence, single dose, change-over trial with oral administration under fasting conditions separated by a washout period of at least 72 hours. Fifty-four healthy participants of both sexes (27 male, 27 female) are intended to be randomized to obtain 42 evaluable participants. The investigational products will be administered in fasted state as single oral doses of 500 mg paracetamol tablet. 1 tablet of test and 1 film-coated tablet of reference 1 and 1 film-coated tablet of reference 2 will be administered in a cross-over manner. Blood sampling will be performed over 24-hour post dose in order to characterize pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the participants participating in the clinical trial.
* Sex: male/female.
* Age: 18 to 55 years (including)
* Body-mass index (BMI): more than or equal to (>=)18.5 kilogram per meter square (kg/m^2) and less than or equal to (<=) 30.0 kg/m^2.
* Body weight: >= 50.0 kg for males and >= 45.0 kg for females.
* Good state of health.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 7 days after the last dose of assigned treatment.
* Non-smoker or ex-smoker for at least 3 months (including non-nicotine vapers, nicotine chewing gum or pouches or nicotine replacement therapy).

Exclusion Criteria:

* Safety Concerns

  1. Existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient.
  2. Existing renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient.
  3. Current evidence of ongoing hepatic disease or impaired hepatic function at screening. A participant will be excluded if more than one of the following lab value deviations are found: 1) Aspartate aminotransferase (AST) (>= 1.2 upper limit of normal [ULN]), Alanine transaminase (ALT) (>= 1.2 ULN), 2) Gamma-glutamyl transferase (GGT) (>= 1.2 ULN), Alkaline phosphatase (ALP) (>= 1.2 ULN), 3) total bilirubin (greater than [>] 2.00 milligrams per deciliter (mg/dL), except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) or creatine kinase (>= 3 ULN), and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 micromole per liter [μmol/l] ULN). A single deviation from the above values is acceptable and will not exclude the candidate, unless specifically advised by the investigator.
  4. Existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient.
  5. History of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders.
  6. History or clinical evidence at screening of pancreatic injury or pancreatitis.
  7. History of inflammatory bowel disease or gastrointestinal bleeding including peptic ulcers.
  8. Diagnosis of systemic lupus erythematosus, thyroid diseases, secondary Raynaud's syndrome; known hyperkalemia.
  9. Evidence of urinary obstruction (example, due to benign prostate hyperplasia) or difficulty in voiding at screening.
  10. Status of glutathione depletion (eating disorder, cystic fibrosis, human immunodeficiency virus [HIV] infection, starvation, cachexia) due to metabolic deficiencies.
  11. Oral surgery within 4 weeks of dosing, dental work or extractions within 2 weeks of dosing, or presence of any clinically significant (as determined by the principal investigator or designee) oral pathology including lesions, sores or inflammation.
  12. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling or gastric banding (note: this is not applicable for minor abdominal surgery without significant tissue resection, example, appendectomy and herniorrhaphy).
  13. Participants, who report a frequent occurrence of migraine attacks.
  14. Acute or chronic diseases which may interfere with the pharmacokinetics of the investigational medicinal product (IMP).
  15. Clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
  16. History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine (> 1.43 mg/dL) or blood urea nitrogen (BUN) (>= 35 mg/dL) or the presence of clinically significant abnormal urinary constituents (example, albuminuria).
  17. Systolic blood pressure less than (<) 90 or > 139 millimeter of mercury (mmHg).
  18. Diastolic blood pressure < 50 or > 89 mmHg.
  19. Heart rate < 50 beats per minute (bpm) or > 90 bpm.
  20. Corrected QT interval (QTc) interval > 450 milliseconds (ms) for men and > 470 ms for women.
  21. Hemoglobin value < 12.0 grams per deciliter (g/dL) for males and < 11.5 g/dL for females.
  22. Evidence or history of medication overuse headache, or allergic disease to medication within the last 5 years that may increase the risk associated with study participation.
  23. Laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator.
  24. Positive anti-HIV-test (if positive to be verified by western blot), hepatitis B surface antigen (HBs-AG) test and anti-hepatitis B core immunoglobulin M (HBc IgM) or anti-hepatitis C virus (HCV) test.
  25. Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations.
  26. Any history of asthma, urticaria, or other significant allergic diathesis or allergic reaction to any other pain reliever/fever reducer. Participant with uncomplicated seasonal allergic rhinitis can be accepted if expected allergy season is clearly outside enrollment/treatment period.
  27. History of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator.
* Lack of suitability for the clinical trial

  1. History of illegal or legal drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana, codeine) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, any opioid derivatives such as heroin or fentanyl, and amphetamine derivatives) within 3 months prior to screening.
  2. Positive alcohol, cotinine or drug test at screening examination.
  3. History of alcohol abuse in the last 5 years or regular intake of alcoholic food or beverages of >= 24 gram (g) pure ethanol for men or >= 12 g pure ethanol for women per day.
  4. Participants who are on a diet which could affect the pharmacokinetics of the active ingredient.
  5. Regular intake of beverages or food containing xanthine derivatives or xanthine-related compounds (example, coffee, tea, caffeine-containing sodas and chocolate), equivalent to >= 500 milligram (mg) xanthine per day.
  6. Performance of strenuous physical exercise (body building, high performance sports) from 2 weeks prior to admission and throughout the entire study.
  7. Participant reports consumption of any drug metabolizing enzyme (example, Cytochrome P450 3A4 (CYP3A4) or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (example, broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort and so on) within 2 weeks prior to admission to the unit.
  8. Use of any systemic or topical medication (including over the counter [OTC] medications, herbal remedies, cannabidiol cosmetics and any anticholinergic medicines or other medicines that may cause dry mouth) within 2 weeks or within less than 10 times the elimination half-life of the respective drug (whichever is longer) before first scheduled study drug administration, or is anticipated to require any concomitant medication during that period or at any time throughout the study.
  9. Any history of long-term treatment with carbamazepine, phenobarbitone, phenytoin, primidone, rifampicin, St John's Wort or other drugs that induce liver enzymes.
  10. Any vaccination, including Coronavirus disease (COVID)-19 vaccine, within 14 days prior to the first dose.
  11. Donation of plasma within 7 days prior to dosing or donation or loss of 500 milliliter (mL) or more of whole blood within 8 weeks prior to dosing.
  12. Participation in a clinical trial in which they have tried an IMP, a medical device or a marketed medicinal product during the last 6 months prior to individual enrolment of the participant.
  13. Simultaneous participation in another clinical trial with active ingredients, medical devices or marketed medicinal products.
* For female participants with childbearing potential only

  1. Positive pregnancy test at screening examination.
  2. Pregnant or lactating women.
  3. Female participants who do not agree to apply highly effective contraceptive methods.
* Administrative reasons

  1. Close affiliation with the sponsor or the investigational site; example, a close relative of the investigator, dependent person (example, employee of or student at the investigational site), employee of the sponsor or affiliates.
  2. Participants who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) for Paracetamol ODT (Test) Versus (Vs) Paracetamol (Alvedon Film-coated Tablet) (Reference 1) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  Cmax is defined as maximum observed post-dose plasma concentration for paracetamol. Blood samples will be collected at indicated timepoints for the analysis of Cmax. Pharmacokinetic (PK) parameters will be determined by non-compartmental analysis.
Area Under the Concentration Versus Time Curve from Dosing Time to the Last Measurement Time Point (AUC0-tlast) for Paracetamol ODT (Test) Vs Paracetamol (Alvedon Film-coated Tablet) (Reference 1) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUC0-tlast is defined as area under the concentration Vs time curve from dosing time to the last measurement time point with a concentration value above the lower limit of quantitation, calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations). Blood samples will be collected at indicated timepoints for the analysis of AUC0-tlast. PK parameters will be determined by non-compartmental analysis.
Time to Reach Maximum Concentration (tmax) for Paracetamol ODT (Test) Vs Paracetamol (Alvedon Film-coated Tablet) (Reference 1) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  Blood samples will be collected at indicated timepoints for the analysis of tmax. PK parameters will be determined by non-compartmental analysis.
Cmax for Paracetamol ODT (Test) Vs Paracetamol (Pandol Film-coated Tablet) (Reference 2) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  Cmax is defined as maximum observed post-dose plasma concentration for paracetamol. Blood samples will be collected at indicated timepoints for the analysis of Cmax. PK parameters will be determined by non-compartmental analysis.
AUC0-tlast for Paracetamol ODT (Test) Vs Paracetamol (Pandol Film-coated Tablet) (Reference 2) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUC0-tlast is defined as area under the concentration Vs time curve from dosing time to the last measurement time point with a concentration value above the lower limit of quantitation, calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations. Blood samples will be collected at indicated timepoints for the analysis of AUC0-tlast). PK parameters will be determined by non-compartmental analysis.
tmax for Paracetamol ODT (Test) Vs Paracetamol (Pandol Film-coated Tablet) (Reference 2) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  Blood samples will be collected at indicated timepoints for the analysis of tmax. PK parameters will be determined by non-compartmental analysis.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve Calculated From Time Zero to Infinity [AUC (0-inf)] for Paracetamol ODT (Test) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUC (0-inf)= AUC0-tlast + AUCexpol, where AUCexpol = Clast/Lz, where Clast is observed concentration at the last time point with a concentration value above the lower limit of quantitation, directly taken from measured concentration values and Lz is apparent terminal elimination rate constant determined by log-linear regression; the regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples will be collected at indicated timepoints for the analysis of AUC (0-inf). PK parameters will be determined by non-compartmental analysis.
AUC (0-inf) for Paracetamol (Alvedon Film-coated Tablet) (Reference 1) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUC (0-inf)= AUC0-tlast + AUCexpol, where AUCexpol = Clast/Lz, where Clast is observed concentration at the last time point with a concentration value above the lower limit of quantitation, directly taken from measured concentration values and Lz is apparent terminal elimination rate constant determined by log-linear regression; the regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples will be collected at indicated timepoints for the analysis of AUC (0-inf). PK parameters will be determined by non-compartmental analysis.
AUC (0-inf) for Paracetamol (Pandol Film-coated Tablet) (Reference 2) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUC (0-inf)= AUC0-tlast + AUCexpol, where AUCexpol = Clast/Lz, where Clast is observed concentration at the last time point with a concentration value above the lower limit of quantitation, directly taken from measured concentration values and Lz is apparent terminal elimination rate constant determined by log-linear regression; the regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples will be collected at indicated timepoints for the analysis of AUC (0-inf). PK parameters will be determined by non-compartmental analysis.
AUCexpol% for Paracetamol ODT (Test) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUCexpol%= AUCexpol*100/AUC0-inf, where AUCexpol = Clast/Lz. Blood samples will be collected at indicated timepoints for the analysis of AUCexpol%. PK parameters will be determined by non-compartmental analysis.
AUCexpol% for Paracetamol (Alvedon Film-coated Tablet) (Reference 1) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUCexpol%= AUCexpol*100/AUC0-inf, where AUCexpol = Clast/Lz. Blood samples will be collected at indicated timepoints for the analysis of AUCexpol%. PK parameters will be determined by non-compartmental analysis.
AUCexpol% for Paracetamol (Pandol Film-coated Tablet) (Reference 2) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  AUCexpol%= AUCexpol*100/AUC0-inf, where AUCexpol = Clast/Lz. Blood samples will be collected at indicated timepoints for the analysis of AUCexpol%. PK parameters will be determined by non-compartmental analysis.
Apparent Terminal Elimination Rate Constant Determined by Log-linear Regression (Lz) for Paracetamol ODT (Test) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  Lz is an apparent terminal elimination rate constant determined by log-linear regression; the regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples will be collected at indicated timepoints for the analysis of Lz. PK parameters will be determined by non-compartmental analysis.
Lz for Paracetamol (Alvedon Film-coated Tablet) (Reference 1) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  Lz is an apparent terminal elimination rate constant determined by log-linear regression; the regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples will be collected at indicated timepoints for the analysis of Lz. PK parameters will be determined by non-compartmental analysis.
Lz for Paracetamol (Pandol Film-coated Tablet) (Reference 2) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  Lz is an apparent terminal elimination rate constant determined by log-linear regression; the regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples will be collected at indicated timepoints for the analysis of Lz. PK parameters will be determined by non-compartmental analysis.
Apparent Terminal Elimination Half-life (t1/2) for Paracetamol ODT (Test) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  t1/2 = ln(2) / Lz. Blood samples will be collected at indicated timepoints for the analysis of t1/2. PK parameters will be determined by non-compartmental analysis.
t1/2 for Paracetamol (Alvedon Film-coated Tablet) (Reference 1) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  t1/2 = ln(2) / Lz. Blood samples will be collected at indicated timepoints for the analysis of t1/2. PK parameters will be determined by non-compartmental analysis.
t1/2 for Paracetamol (Pandol Film-coated Tablet) (Reference 2) | Within one hour prior to dosing, at 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 75, 90, 120, 150, 180 minutes and at 4, 5, 6, 8, 10, 12, 14, 16 and 24 hours following dosing in each treatment period
  t1/2 = ln(2) / Lz. Blood samples will be collected at indicated timepoints for the analysis of t1/2. PK parameters will be determined by non-compartmental analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- SocraTec R&D GmbH, Erfurt, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trialregister@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.